CLINICAL TRIAL: NCT02732132
Title: A Comparison of the Sedation With Intermittent Bolus Midazolam-Ketamine Versus Intermittent Bolus Propofol-Fentanyl During Endoscopy in Children: Randomized Trial
Brief Title: A Comparison of the Sedation During Endoscopy in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ulas Emre Akbulut, Medical Doctor, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2015/18
Record Dates: First submitted 2016-03-23; First posted 2016-04-08 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2016-04

CONDITIONS: Failed Moderate Sedation During Procedure
MeSH Terms: interventions — Ketamine; Midazolam; Propofol; Fentanyl

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine and Midazolam (Active Comparator): ketamine 1 mg/kg midazolam 0.1 mg/kg
  Interventions: Drug: Ketamine and Midazolam
- Propofol and Fentanyl (Experimental): propofol 1 mg/kg fentanyl 1 mcg/kg
  Interventions: Drug: Propofol and Fentanyl

INTERVENTIONS:
Drug: Ketamine and Midazolam — This group was injected intravenous midazolam 0.1 mg/kg (maximum 4 mg), two minutes later, ketamine 1 mg/kg was given intravenously before the start of endoscopy.
  Other Names: Ketalar (Ketamin, Pfizer) and Dormicum (Midazolam, Roche)
  Arms: Ketamine and Midazolam
Drug: Propofol and Fentanyl — This group was injected intravenous fentanyl 1 mcg/kg, and two minutes later, propofol 1 mg/kg was given intravenously before the start of endoscopy.
  Other Names: Propofol Lipuro (Propofol, B-Braun) Fentanyl (Fentanyl, J&J)
  Arms: Propofol and Fentanyl

SUMMARY:
The primary aim of this study was to investigate the efficiency and safety of midazolam plus ketamine versus fentanyl plus propofol administered to children undergoing UGE and to determine the most appropriate sedation protocol.

DETAILED DESCRIPTION:
The patients were given a spray of lidocaine 10% as a topical pharyngeal anaesthesia before sedation. Intravenous midazolam bolus dose 0.1 mg/kg (maximum 4 mg) was administered to Group A. Two minutes later, ketamine bolus dose 1 mg/kg was given intravenously. Patient responses to verbal and tactile stimuli were evaluated two minutes after ketamine application. Ketamine 0.5 mg/kg (maximum of 2 mg/kg) was added in two minute intervals if adequate sedation was not achieved initially. The endoscopy process was initiated by the endoscopist if there was no response. If the patients were agitated after the procedure started, a ketamine 0.5 mg/kg single dose was applied. Intravenous fentanyl bolus dose 1µg/kg was administered to Group B. Two minutes later, propofol bolus dose 1 mg/kg was given intravenously. Patient responses to verbal and tactile stimuli were evaluated two minutes after propofol application. Propofol 0.5 mg/kg was added in two minute intervals if adequate sedation was not achieved. The endoscopy process was initiated by the endoscopist if there was no response. If the patients were agitated after the procedure started, a propofol 0.5 mg/kg single dose was applied. None of the patients were given an antidote after the process during recovery.

All patients were monitored for peripheral oxygen saturation, heart rate (HR), respiratory rate, and RSS during the procedure. Oxygen (2L/min) by nasal cannula was given to all patients during the procedure. Hypoxia (peripheral oxygen saturation <90% during 60 seconds), apnea, laryngospasm, tachycardia (defined as 30% more than the average heart rate by age), bradycardia (30% less than the average heart rate by age), increase in oral secretions (more than enough to warrant aspiration), flushing, coughing and vomiting were assessed as complications and recorded.

ELIGIBILITY:
Inclusion Criteria:

* All the patients were in ASA (American Society of Anesthesiologists) physical status I or II.

Exclusion Criteria:

* Patients with respiratory tract infections, glaucoma, psychosis, porphyria, hypertension, metabolic or neurologic diseases, increased intracranial pressure and intracranial mass, and patients known to be allergic to the drugs used were excluded from the study.

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 238 (Actual)
Dates: Start 2015-01; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
the effectiveness of sedation | six months
  the effectiviness of midazolam plus ketamine versus fentanyl plus propofol according to a modified Ramsay sedation score

SECONDARY OUTCOMES:
adverse events that are related to study drugs | six months
  number of patients with adverse events that are related to study drugs
procedure time | six months
  procedure time is defined as the time between the insertion of endoscope and removal of endoscope
recovery time | six months
  recovery time is defined as the time from completing the endoscopy to achieving Aldrete score 10 in the recovery unit Aldrete score

IPD SHARING:
Plan to Share IPD: No